CLINICAL TRIAL: NCT02486458
Title: Retention of Fluoride Formed on Enamel by Fluoride Gel or Varnish Application and Its Release to Dental Biofilm Fluid - in Vivo Study
Brief Title: Long-term Release of Fluoride Formed on Enamel by Fluoride Gel or Varnish to Biofilm Fluid
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Livia Maria Andaló Tenuta, DDS, MSc, PhD, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FOPBioq005
Record Dates: First submitted 2015-05-26; First posted 2015-07-01 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Dental Caries
Keywords: Fluoride; Biofilm fluid; Calcium fluoride; Topical
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Negative control (No Intervention): No treatment will be applied
- Varnish 4 h (Experimental): Fluoride varnish will be applied on teeth and removed after 4 hours
  Interventions: Drug: 5% sodium fluoride varnish
- Varnish 24 h (Experimental): Fluoride varnish will be applied on teeth and removed after 24 hours
  Interventions: Drug: 5% sodium fluoride varnish
- Fluoride Gel (Experimental): Fluoride gell will be applied on teeth and removed after 4 minutes
  Interventions: Drug: 1.23% sodium fluoride acidic gel

INTERVENTIONS:
Drug: 5% sodium fluoride varnish — Fluoride varnish containing 22,600 ppm F, as NaF, in a neutral base
  Arms: Varnish 24 h; Varnish 4 h
Drug: 1.23% sodium fluoride acidic gel — Fluoride gel containing 12,300 ppm F (as NaF) in an acidic pH (by addition of phosphoric acid)
  Arms: Fluoride Gel

SUMMARY:
The anticaries effect of professional fluoride application has been associated with the formation of calcium fluoride-like products ("CaF2") on dental surface, which may function as a slow release fluoride reservoir. Among professional fluoride products, fluoride gel and varnish are the most important, and have different soluble fluoride concentrations, pHs and vehicles. Although the concentration of fluoride formed on enamel after the use of both is similar, the retention of these reaction products is unknown. Also, it is unknown the capacity of these reservoirs to enhance dental biofilm fluid with fluoride. Moreover, the effect of the varnish application time on these parameters is unknown. Therefore, the aim of this study is to compare the capacity of fluoride gel and varnish to form fluoride reservoirs on enamel and increase dental biofilm fluid fluoride concentration with time. Rapid biofilm-forming individuals will be selected to participate and divided into 4 experimental groups: 1. Negative control: no treatment; 2. Varnish 4 hours: fluoride varnish will be applied and kept on teeth for 4 hours; 3. Varnish 24 h: fluoride varnish will be applied on teeth and kept for 24 h; and 4. Gel: Fluoride gel will be applied on teeth. Microbiopsies of enamel will be obtained by a microbiospy technique to assess fluoride concentration before, 7 and 28 days after the treatments. Dental biofilm will be collected before and 3, 7, 14 and 28 days after treatments. Fluoride concentration on enamel and in the biofilm fluid will be determined by an ion-specific electrode. Data will be analyzed statistically comparing the groups and collection times.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Good oral health
* At least 5 teeth in each hemiarch
* All 4 superior incisors in the mouth
* Rapid biofilm forming

Exclusion Criteria:

* Pregnancy
* Intake of medication that reduces salivary flow
* Chronic diseases
* Smokers
* Orthodontic appliances
* Dental prosthesis
* Allergy to fluoride varnish components

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in fluoride concentration in enamel days after fluoride application | Up to 28 days
Change in fluoride concentration in dental biofilm fluid days after fluoride application | Up to 28 days

SECONDARY OUTCOMES:
Change in fluoride concentration in whole biofilm days after fluoride application | Up to 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Unochapecó, Chapecó, Santa Catarina, Brazil